CLINICAL TRIAL: NCT05485181
Title: Validating Promoted Spiritual Experience: A Pilot Study
Brief Title: Validating Promoted Spiritual Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Damon House (Unknown); Rutgers Brain Health Institute (Unknown)
Responsible Party: Principal Investigator, John Calvin Chatlos, MD, Medical Director SATS, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro2022000889
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Addiction; Psychiatric Disorder
Keywords: spirituality; neuroimaging; CBT; self-worth; dignity
MeSH Terms: conditions — Behavior, Addictive; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Two cohorts of 8 subjects each will receive psychological assessments initially.
  First cohort will have brain scan followed by 9 week intervention and post-intervention repeat scan and repeat assessments.
  2nd cohort serves as its own control, will receive repeat assessments and brain scan after Cohort 1 is done, and again after 9 week intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 8 subjects get psychological assessments and fMRI brain scan followed by 9 week psychotherapeutic intervention. With intervention completion, psychological assessments and fMRI scan are repeated.
  Interventions: Behavioral: Spiritual Intervention
- Cohort 2 (Active Comparator): 8 subjects get psychological assessments at same time as Cohort 1, but do not receive the intervention at that time - serving as control group.
  When Cohort 1 is completed, Cohort 2 will repeat psychological assessments, receive fMRI scan, then receive same 9 week intervention as Cohort 1, followed by repeat psychological assessments and fMRI scan.
  Interventions: Behavioral: Spiritual Intervention

INTERVENTIONS:
Behavioral: Spiritual Intervention — The Intervention is a CBT- based psychotherapeutic process that occurs in a group setting with two cohorts of 8 subjects each. It will occur in an introductory 3-hour session followed by 9 weekly 1 ½ hour sessions. In this process, self-worth (self-confidence, self-esteem, self-competence) and dignity (reason, compassion, courage) as operationally defined are strengthened through an interpersonal, psychological process including mindful self-awareness training, attitude transformation with self-compassion, forgiveness, and self-acceptance, and opens to a new level of awareness. This awareness opens to spiritual / numinous features of connectedness, vitality, wholeness, meaning, and serenity that are predicted to be associated with greater well-being and relief of anxiety and depression symptoms.

SUMMARY:
This pilot study of 16 patients will demonstrate a specific psychologically focused intervention to affect a spiritual aspect of psychological health and will measure (1) its effects on general distress, depression, anxiety and well-being; (2) healing and psychological impact beyond that accounted by usual personality factors; (3) its effect in correlation to measures of spirituality; (4) with neuroimaging, possible biological changes associated with this intervention.

A. Objectives

1. Pilot a psychological intervention that impacts a "spiritual" level.
2. Measure efficacy improving well-being beyond explanation by usual personality factors.
3. Identify biological changes with neuroimaging.

B. Hypotheses / Research Question(s) Studies demonstrate a healing effect beyond usual psychological and medical health to include a "spiritual" aspect with added experience of wholeness and well-being. Benefits are beyond just symptom relief but methods to achieve this are not well-defined. This study will provide a specific intervention and measure psychological and neuroimaging effects of the intervention.

Hypotheses of Specific Results (see Study Instruments below)

1. DASS-21-shows significant decrease in depression, anxiety and overall stress.
2. PCL-5 - shows decrease 5-10 points (5 points=response, 10 points=clinically meaningful).
3. NIH-HEALS - shows significant increase overall and in all 3 factors.
4. WEMWBS - shows increase of greater than 3 points, considered "meaningful change."
5. Contingencies of Self-Worth Scale-shows significant global increase, positively correlated with increase in Mysticism Scale scores with post-intervention total above standardized mean.
6. A relevant portion of outcome improvement on DASS-21, NIH-HEALS, and ASPIRES will NOT be accountable by personality factors measured by NEO-FFI-3.
7. ASPIRES-shows significant increase in transcendence, no change in religious sentiments.
8. Neuroimaging-shows reduced activity in SPL, TPJ, MPFC, and IPL (see Research Significance).

DETAILED DESCRIPTION:
Following IRB approval, recruit 16 patients from a male residential addiction treatment program for a 10-session intervention. 8 subjects will be given pre and post intervention psychological assessments and pre and post fMRIs. Another 8 subjects will serve as a control group and will receive the pre and post (without intervention) psychological assessments at the same time as the previous group and will then be the next 8 subjects to receive the intervention after completion of the first cohort. They will have MRIs before their intervention and post-intervention, thus serving as their own control group. The behavioral intervention occurs with a beginning 3 hour group introduction done by Dr. Chatlos followed by 9 weekly 1 ½ hour group sessions. The subjects' intervention will be recorded for further manual development.

The Intervention is a CBT- based psychotherapeutic process that occurs in a group setting with two cohorts of 8 subjects each. It will occur in an introductory 3-hour session followed by 9 weekly 1 ½ hour sessions. In this process, self-worth (self-confidence, self-esteem, self-competence) and dignity (reason, compassion, courage) as operationally defined are strengthened through an interpersonal, psychological process including mindful self-awareness training, attitude transformation with self-compassion, forgiveness, and self-acceptance, and opens to a new level of awareness. This awareness opens to spiritual / numinous features of connectedness, vitality, wholeness, meaning, and serenity that are predicted to be associated with greater well-being and relief of anxiety and depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Recently admitted (within 3 months) male patients of a residential addiction treatment program that has a 6 month average duration.
* Age 21 or older.
* Volunteer for the study after a brief introduction.

Exclusion Criteria:

* No psychosis, no suicidal ideation or psychiatric hospitalization in past 3 months.
* Usual MRI Exclusionary Criteria detailed in IRB

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
NIH-HEALS | 12 weeks
  (NIH-Healing Experience of All Life Stressors) (Ameli et al, 2018): 35-item Likert scale strongly disagree 1 to 5 strongly agree. 3 factor structure:connection (range 10-50), reflection (range 14-70 & trust & acceptance (range 11-55. Total range: 35-175. Higher score is better. Expected change in all 3 scales.
fMRI Scan | 12 weeks
  fMRI Neuroimaging-will show change in activity in MPFC, SPL, TPJ, and IPL

SECONDARY OUTCOMES:
Depression, Anxiety, Stress | 12 weeks
  DASS-21 (Depression, Anxiety, and Stress Scale) (Henry, 2005): 21-item Likert scale Never 0 to 3 Almost always, lower is better. Range each scale: 0-21. Expected change in depression, anxiety and overall stress scales.
Well-Being | 12 weeks
  WEMWBS (Warwick-Edinburgh Mental Wellbeing Scale) (Warwick, 2018) measures psychological well-being; 14-item Likert scale None of the time 1 to 5 All of the time. Range: 14-70, higher is better. Expected change in overall score.
Transcendence | 12 weeks
  ASPIRES (Assessment of Spirituality and Religious Sentiments) (Piedmont, 2009): 35-item Likert scale strongly agree 1 to 5 strongly disagree. 2 main factors- religious sentiments (RS) (Range 12-60) and spiritual transcendence(ST) (Range:23-115) . Expected outcome is change in ST scale only.
Personally Independent Effects | 12 weeks
  NEO-FFI-3 (NEO-Five Factor Inventory) (McRae, 2007): 60-item yes/no response FFM (Five Factor Model) of personality- Neuroticism, Extraversion, Openness to experience, Agreeableness, and Conscientiousness.Range: 0-12, higher is greater. No expected change, used for comparison.
PTSD | 12 weeks
  PTSD Checklist for DSM-5(PCL-5) (Blevins, 2015): 20-item Likert scale Not at all 0 to 4 Extremely. Range: 14-70, lower is better. Expected outcome is change in overall score.

OTHER OUTCOMES:
Spirituality - Mysticism Measure | 12 weeks
  Mysticism Scale-Research Form D (Hood,1975): 32-item Likert scale 5-point Strongly Agree to Strongly Disagree. Range: 32-160 toal. Eight factors: ego quality, unifying quality, inner subjective quality, temporal/spatial quality, noetic auality, positive affect, religious quality. Expected outcome is a change in all factors.
Theory Validity Self-Worth | 12 weeks
  Contingencies of Self-Worth Scale (Crocker, 2003): 35-item Likert scale Strongly Agree 1 to 7 Strongly Disagree, higher is better. Measures global self-worth (Range: 30-210) and 6 factors (Range:5-35) with 6 factors. Expected outcome is change in global self-worth total.
NMI | 12 weeks
  Numinous Motivation Inventory (Piedmont 2017) 22-item Likert scale Strongly Disagree 1 to 5 Strongly Agree, Range: 22-110, higher is better. Expected outcome is change of total score.
Human Spirituality Scale | 12 weeks
  HHS (Wheat 1991) 21-item Likert scale 5 point, end ponts vary. Range: 21-105, lower is greater. Expected outcome is change of total score.

CONTACTS AND LOCATIONS:
Overall Officials: Kasia Bieszczad, PhD, Principal Investigator — Rutgers University - Dept Psychology; Nina Cooperman, PhD, Principal Investigator — Rutgers University - Dept Psychiatry
Locations (1):
- Rutgers - The State University of New Jersey, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data that underlie the results of the study after de-identification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 3 months after published paper to 2 years.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Miller L, Balodis IM, McClintock CH, Xu J, Lacadie CM, Sinha R, Potenza MN. Neural Correlates of Personalized Spiritual Experiences. Cereb Cortex. 2019 Jun 1;29(6):2331-2338. doi: 10.1093/cercor/bhy102. PMID 29846531
- See also: Chatlos, J. Framework of Spirituality — https://doi.org/10.1111/zygo.12670